CLINICAL TRIAL: NCT01685060
Title: A Phase II, Multicenter, Single-arm Study of Oral LDK378 in Adult Patients With ALK-activated Non-small Cell Lung Cancer Previously Treated With Chemotherapy and Crizotinib
Brief Title: LDK378 in Adult Patients With ALK-activated NSCLC Previously Treated With Chemotherapy and Crizotinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDK378A2201; 2012-003432-24 (EudraCT Number)
Record Dates: First submitted 2012-09-04; First posted 2012-09-13 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; ALK; LDK378; Ceritinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LDK378 (Experimental): Patients treated with ceritinib/LDK378 750 mg once-daily, fasted
  Interventions: Drug: LDK378

INTERVENTIONS:
Drug: LDK378 — Ceritinib/LDK378 was supplied as 150 mg hard gelatin capsules and were administered orally, once-daily at a dose of 750 mg on a continuous dosing schedule (5 x 150 mg capsules).
  Other Names: Ceritinib

SUMMARY:
A single-arm, open-label, multicenter, phase II study. Treatment with LDK378 750 mg qd continued until the patient experienced unacceptable toxicity that precluded further treatment, discontinued treatment at the discretion of the investigator or patient, started a new anti-cancer therapy and/or died. LDK378 could be continued beyond RECIST-defined progressive disease (PD) as assessed by the investigator if, in the judgment of the investigator, there was evidence of clinical benefit. In these patients tumor assessment would continue as per the schedule of assessments until treatment with LDK378 was permanently discontinued. Patients who discontinued the study medication in the absence of progression continued to be followed for tumor assessment until the time of PD as assessed by the investigator

ELIGIBILITY:
Inclusion critieria:

* Histologically or cytologically confirmed diagnosis of stage IIIB or IV NSCLC that carries an ALK rearrangement, as per the FDA-approved FISH assay (Abbott Molecular Inc.).
* Age 18 years or older at the time of informed consent.
* Patients must have NSCLC that has progressed during therapy with crizotinib or within 30 days of the last dose
* Patients must have received 1-3 lines of cytotoxic chemotherapy (of which 1 must have been a platinum doublet) to treat their locally advanced or metastatic NSCLC
* Patients must have a tumor tissue sample available, collected either at the time of diagnosis of NSCLC or any time since.
* Patients must have recovered from all toxicities related to prior anticancer therapies to grade ≤ 2, except for patients with grade 2 nausea/vomiting and/or grade 2 diarrhea despite optimal supportive therapy who will not be allowed to participate in the study.

Exclusion criteria:

* Patients with known hypersensitivity to any of the excipients of LDK378.
* Patients with symptomatic central nervous system (CNS) metastases who are neurologically unstable or have required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms.
* History of carcinomatous meningitis.
* Presence or history of a malignant disease other than NSCLC that has been diagnosed and/or required therapy within the past 3 years.
* Clinically significant, uncontrolled heart disease
* Systemic anti-cancer therapy given after the last dose of crizotinib and prior to starting study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-11-26 (Actual); Primary Completion 2016-03-29 (Actual); Study Completion 2016-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (50):
- United States (17):
  - Highlands Oncology Group Dept of Highlands Oncology Grp, Fayetteville, Arkansas
  - City of Hope National Medical Center Dept of Oncology 2, Duarte, California
  - University of California at Los Angeles Reg-5, Los Angeles, California
  - University of California at San Diego, Moores Cancer Ctr SC, San Diego, California
  - Stanford University Medical Center Stanford Cancer Center(2), Stanford, California
  - University of Colorado Hospital SC, Aurora, Colorado
  - Emory University School of Medicine/Winship Cancer Institute Dept of Oncology, Atlanta, Georgia
  - University of Chicago Medical Center SC, Chicago, Illinois
  - University of Kansas Cancer Center DeptofUofKansas CancerCenter-2, Kansas City, Kansas
  - Cancer Center of Kansas Dept of CCK, Wichita, Kansas
  - Maryland Oncology Hematology, P.A. SC, Rockville, Maryland
  - Massachusetts General Hospital Mass General, Boston, Massachusetts
  - Levine Cancer Institute SC 1, Charlotte, North Carolina
  - Sarah Cannon Research Institute Drug Ship - 4, Nashville, Tennessee
  - U of TX Southwestern Medical Center - SimmonsCompCancerCtr Clinical Research Office, Dallas, Texas
  - Seattle Cancer Care Alliance SC-1, Seattle, Washington
  - University of Wisconsin Univ Wisc 2, Madison, Wisconsin
- Canada (3):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Oshawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
- France (2):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
- Germany (2):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Heidelberg
- Novartis Investigative Site, Hong Kong, Hong Kong
- Italy (6):
  - Novartis Investigative Site, Avellino, AV
  - Novartis Investigative Site, Livorno, LI
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Parma, PR
- Japan (9):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Akashi, Hyōgo
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Sayama, Osaka
  - Novartis Investigative Site, Sunto-gun, Shizuoka
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Koto, Tokyo
  - Novartis Investigative Site, Fukuoka
- Netherlands (3):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Maastricht
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, Korea, South Korea
- Spain (4):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, London, United Kingdom

REFERENCES:
- [Derived] Hida T, Satouchi M, Nakagawa K, Seto T, Matsumoto S, Kiura K, Nokihara H, Murakami H, Tokushige K, Hatano B, Nishio M. Ceritinib in patients with advanced, crizotinib-treated, anaplastic lymphoma kinase-rearranged NSCLC: Japanese subset. Jpn J Clin Oncol. 2017 Jul 1;47(7):618-624. doi: 10.1093/jjco/hyx045. PMID 28369553
- [Derived] Crino L, Ahn MJ, De Marinis F, Groen HJ, Wakelee H, Hida T, Mok T, Spigel D, Felip E, Nishio M, Scagliotti G, Branle F, Emeremni C, Quadrigli M, Zhang J, Shaw AT. Multicenter Phase II Study of Whole-Body and Intracranial Activity With Ceritinib in Patients With ALK-Rearranged Non-Small-Cell Lung Cancer Previously Treated With Chemotherapy and Crizotinib: Results From ASCEND-2. J Clin Oncol. 2016 Aug 20;34(24):2866-73. doi: 10.1200/JCO.2015.65.5936. Epub 2016 Jul 18. PMID 27432917

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Approximately 137 patients were planned to be enrolled. A total of 140 patients were enrolled and treated with ceritinib.
Groups:
- LDK378 750mg: Patients treated with ceritinib/LDK378 750 mg once-daily, fasted.
Period: Overall Study
Arm/Group | LDK378 750mg
Started | 140
Entered Post-treatment Efficacy f/u | 7
Entered Survival Follow up | 98
Discontinued From Study | 35
Completed | 0
Not Completed | 140
Not completed — Rollover patients | 16
Not completed — Adverse Event | 12
Not completed — Progressive disease | 69
Not completed — Physician Decision | 14
Not completed — Subject/guardian decision | 20
Not completed — Lost to Follow-up | 1
Not completed — Death | 8

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) consisted of all patients who received at least one dose of ceritinib.
Arm/Group | LDK378 750mg
Number analyzed (Participants) | 140
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.2 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 70

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) to LDK378 Per Investigator Assessment
Description: ORR per RECIST 1.1 calculated as the percentage of patients with a best overall confirmed response defined as complete response or partial response (CR+PR) as assessed by investigator. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm 1. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: 6 cycles of 28 days up to 24 weeks
Population: Full Analysis Set (FAS) consisted of all patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378 750mg
Number analyzed (Participants) | 140
Percentage of participants | 40.7 [32.5 to 49.3]

2. Secondary Outcome: ORR Per Blinded Independent Review Committee (BIRC) Assessment
Description: ORR (CR+PR) by BIRC is calculated as the percentage of patients with a best overall confirmed response defined as complete response or partial response (CR+PR) as assessed by BIRC. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm 1. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: 6 cycles of 28 days up to 24 weeks
Population: The Full Analysis Set (FAS) consists of all patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378 750mg
Number analyzed (Participants) | 140
Percentage of participants | 35.7 [27.8 to 44.2]

3. Secondary Outcome: Duration of Response (DOR) by Investigator
Description: DOR, calculated as the time from the date of the first confirmed CR or PR to the first documented progression or death due to any cause, by investigator. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm 1. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: 6 cycles of 28 days up to 24 weeks
Population: Full Analysis Set (FAS) consisted of all patients who received at least one dose of ceritinib. Only patients with confirmed complete response/partial response (CR/PR) per Investigator were included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDK378 750mg
Number analyzed (Participants) | 57
Months | 10.6 [7.4 to 14.7]

4. Secondary Outcome: Duration of Response (DOR) by BIRC
Description: DOR, calculated as the time from the date of the first documented CR or PR to the first documented progression or death due to underlying cancer, by BIRC (Blinded Imaging Review Committee). CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm 1. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: 6 cycles of 28 days up to 24 weeks
Population: Full Analysis Set (FAS) consisted of all patients who received at least one dose of ceritinib. Only patients with confirmed complete response/partial response (CR/PR) per BIRC were included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDK378 750mg
Number analyzed (Participants) | 50
Months | 12.9 [9.3 to 18.4]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was calculated as the percentage of patients with best overall response of CR, PR, SD, or non-CR non-PD (NCRNPD), per RECIST 1.1 by investigator. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm 1. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD. Non-CR/Non-PD (NCRNPD): refers to best overall responses that are neither CR nor PD per RECIST 1.1 criteria for patients with non-measurable disease only at baseline.
Time Frame: 6 cycles of 28 days up to 24 weeks
Population: Full Analysis Set (FAS) consisted of all patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378 750mg
Number analyzed (Participants) | 140
Percentage of participants
  DCR per Investigator | 76.4 [68.5 to 83.2]
  DCR per BIRC | 80.0 [72.4 to 86.3]

6. Secondary Outcome: Time to Response (TTR) Per Investigator
Description: TTR is the time from date of start of treatment to the first CR or PR observed which were confirmed afterwards.
Time Frame: 6 cycles of 28 days up to 24 weeks
Population: The Full Analysis Set (FAS) consists of all patients who received at least one dose of ceritinib. Only patients with confirmed complete response/partial response (CR/PR) were included in this analysis.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | LDK378 750mg
Number analyzed (Participants) | 57
Months | 3.0 (3.54) [1.6 to 18.7]

7. Secondary Outcome: Time to Response (TTR) Per BIRC
Description: TTR is the time from date of start of treatment to the first CR or PR observed which are confirmed afterwards.
Time Frame: 6 cycles of 28 days up to 24 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | LDK378 750mg
Number analyzed (Participants) | 50
Months | 2.2 (1.44) [1.6 to 10.9]

8. Secondary Outcome: Progression-free Survival (PFS) Per Investigator
Description: PFS, defined as the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient had no event or when the patient received any further anticancer therapy in the absence of disease progression, progression-free survival was censored at the date of last adequate tumor assessment.
Time Frame: 6 cycles of 28 days up to 24 weeks
Population: The Full Analysis Set (FAS) consists of all patients who received at least one dose of ceritinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LDK378 750mg
Number analyzed (Participants) | 140
months | 5.8 [5.4 to 7.6]

9. Secondary Outcome: Progression-free Survival (PFS) Per BIRC
Description: as for outcome 8
Time Frame: 6 cycles of 28 days up to 24 weeks
Population: The Full Analysis Set (FAS) consists of all patients who received at least one dose of ceritinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LDK378 750mg
Number analyzed (Participants) | 140
months | 7.4 [5.6 to 10.9]

10. Secondary Outcome: Overall Intracranial Response Rate (OIRR) Per Investigator
Description: OIRR calculated as the ORR (CR+PR) of lesions in the brain for patients who had measureable disease in the brain at baseline.
Time Frame: 6 cycles of 28 days up to 24 weeks
Population: The Full Analysis Set (FAS) consists of all patients who received at least one dose of ceritinib. Only patients with measurable disease in brain at baseline selected by Investigator were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378 750mg
Number analyzed (Participants) | 20
Percentage of participants | 45.0 [23.1 to 68.5]

11. Secondary Outcome: Overall Intracranial Response Rate (OIRR) Per BIRC
Description: as for outcome 10
Time Frame: 6 cycles of 28 days up to 24 weeks
Population: The Full Analysis Set (FAS) consists of all patients who received at least one dose of ceritinib. Only patients with measurable disease in brain at baseline selected by BIRC were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378 750mg
Number analyzed (Participants) | 28
Percentage of participants | 35.7 [18.6 to 55.9]

12. Secondary Outcome: Overall Survival (OS)
Description: OS, defined as the time from date of randomization/start of treatment to date of death due to any cause. If a patient was not known to have died, survival was censored at the date of last known date patient alive.
Time Frame: 6 cycles of 28 days up to 24 weeks
Population: Full Analysis Set (FAS) consisted of all patients who received at least one dose of ceritinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDK378 750mg
Number analyzed (Participants) | 140
Months | 15.6 [13.6 to 24.2]

ADVERSE EVENTS:
Time Frame: Timeframe for AE
Description: AE additional description
Groups:
- LDK378 750 mg: Patients treated with ceritinib/LDK378 750 mg once-daily, fasted.
Arm/Group | LDK378 750 mg
Serious Adverse Events (participants affected / at risk) | 67/140
Other Adverse Events (participants affected / at risk) | 139/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDK378 750 mg (N=140)
ANAEMIA (Blood and lymphatic system disorders) | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 2
PERICARDITIS (Cardiac disorders) | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 3
ASCITES (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
DYSPHAGIA (Gastrointestinal disorders) | 1
FAECALOMA (Gastrointestinal disorders) | 1
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1
GASTROINTESTINAL TOXICITY (Gastrointestinal disorders) | 1
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 3
PANCREATITIS (Gastrointestinal disorders) | 2
RETROPERITONEAL FIBROSIS (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 4
ASTHENIA (General disorders) | 3
DISEASE PROGRESSION (General disorders) | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2
MALAISE (General disorders) | 3
NON-CARDIAC CHEST PAIN (General disorders) | 3
PAIN (General disorders) | 2
PYREXIA (General disorders) | 8
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1
HEPATOCELLULAR INJURY (Hepatobiliary disorders) | 1
EMPYEMA (Infections and infestations) | 1
ENTERITIS INFECTIOUS (Infections and infestations) | 1
LUNG INFECTION (Infections and infestations) | 1
MENINGITIS (Infections and infestations) | 1
PLEURAL INFECTION (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 6
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
SEPTIC SHOCK (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 1
VIRAL PERICARDITIS (Infections and infestations) | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1
BLOOD CALCIUM INCREASED (Investigations) | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1
BLOOD CREATININE INCREASED (Investigations) | 2
WEIGHT DECREASED (Investigations) | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 2
DEHYDRATION (Metabolism and nutrition disorders) | 4
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO MENINGES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1
APHASIA (Nervous system disorders) | 2
BRAIN OEDEMA (Nervous system disorders) | 2
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1
DYSARTHRIA (Nervous system disorders) | 1
ENCEPHALOPATHY (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 1
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 1
HYPERAESTHESIA (Nervous system disorders) | 1
LETHARGY (Nervous system disorders) | 1
MOTOR DYSFUNCTION (Nervous system disorders) | 1
PARAESTHESIA (Nervous system disorders) | 1
PARAPARESIS (Nervous system disorders) | 1
SEIZURE (Nervous system disorders) | 4
SENSORY LOSS (Nervous system disorders) | 1
CONFUSIONAL STATE (Psychiatric disorders) | 2
HYDRONEPHROSIS (Renal and urinary disorders) | 1
POLLAKIURIA (Renal and urinary disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 2
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 3
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDK378 750 mg (N=140)
ANAEMIA (Blood and lymphatic system disorders) | 25
ABDOMINAL PAIN (Gastrointestinal disorders) | 45
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 16
CONSTIPATION (Gastrointestinal disorders) | 42
DIARRHOEA (Gastrointestinal disorders) | 115
NAUSEA (Gastrointestinal disorders) | 115
STOMATITIS (Gastrointestinal disorders) | 11
VOMITING (Gastrointestinal disorders) | 92
ASTHENIA (General disorders) | 25
FATIGUE (General disorders) | 54
NON-CARDIAC CHEST PAIN (General disorders) | 25
OEDEMA PERIPHERAL (General disorders) | 19
PYREXIA (General disorders) | 28
NASOPHARYNGITIS (Infections and infestations) | 9
PNEUMONIA (Infections and infestations) | 9
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 18
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 65
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 55
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 23
BLOOD CREATININE INCREASED (Investigations) | 27
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 12
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 26
WEIGHT DECREASED (Investigations) | 48
DECREASED APPETITE (Metabolism and nutrition disorders) | 59
HYPOKALAEMIA (Metabolism and nutrition disorders) | 8
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 9
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 16
BACK PAIN (Musculoskeletal and connective tissue disorders) | 28
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 9
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 14
MYALGIA (Musculoskeletal and connective tissue disorders) | 10
NECK PAIN (Musculoskeletal and connective tissue disorders) | 11
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 14
DIZZINESS (Nervous system disorders) | 15
DYSGEUSIA (Nervous system disorders) | 12
HEADACHE (Nervous system disorders) | 31
PARAESTHESIA (Nervous system disorders) | 8
ANXIETY (Psychiatric disorders) | 11
INSOMNIA (Psychiatric disorders) | 18
COUGH (Respiratory, thoracic and mediastinal disorders) | 33
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 29
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 10
ALOPECIA (Skin and subcutaneous tissue disorders) | 9
DRY SKIN (Skin and subcutaneous tissue disorders) | 10
PRURITUS (Skin and subcutaneous tissue disorders) | 8
RASH (Skin and subcutaneous tissue disorders) | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety